CLINICAL TRIAL: NCT02230917
Title: A Phase IIa Study of Sotatercept on Bone Mass and Turnover in Patients With Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Rebecca Silbermann (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Rebecca Silbermann, Assistant Professor, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IUCRO-0428
Record Dates: First submitted 2014-08-19; First posted 2014-09-03 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ACE-011; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sotatercept (Experimental): Sotatercept 0.2 mg/kg will be administered every 21 days for 12 doses subcutaneously into the upper arm, abdomen or thigh.
  Interventions: Drug: Sotatercept
- Placebo (Placebo Comparator): 0.2 mg/kg of normal saline will be administered subcutaneously in the upper arm, abdomen or thigh for 21 days for 12 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotatercept
  Other Names: ACE-011
  Arms: Sotatercept
Drug: Placebo
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Lytic bone disease continues to be one of the most devastating complications of multiple myeloma (MM) despite recent and dramatic advancements in MM management, and bone lesions persist and can continue to significantly impact a patient's morbidity, even when an individual's myeloma is otherwise under good control. To date, no agent has been shown to have a prolonged bone anabolic response in myeloma.

Preliminary studies treating healthy postmenopausal women with a single dose of sotatercept demonstrated a rapid and sustained increase in serum biochemical markers of bone formation and a decrease in markers of bone resorption. Similarly, the murine analog to sotatercept, RAP-011, increases bone mineral density and strength in murine studies of both normal animals and models of bone loss. We hypothesize that sotatercept will provide an anabolic response for bone in myeloma patients with bone disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years at the time of signing the informed consent form.
2. Documented diagnosis of Multiple Myeloma, currently with complete response (CR) or very good partial response (VGPR) (as defined by IMWG criteria), at least two years after induction therapy or autologous stem cell transplant.
3. Patients must not be receiving anti-Myeloma therapy (including maintenance therapy).
4. Disease response must be confirmed with repeat laboratory studies at least 30 days apart.
5. Radiologic evidence of at least 1 measurable lytic lesion in the arm, pelvis or leg. Completion of two years monthly zoledronic acid therapy.
6. Eastern Cooperative Group (ECOG) performance status 0- 2
7. Creatinine ≤1.5 x upper limit of normal (ULN) or ≥40 mL/min
8. Total bilirubin ≤ 3.0 mg/dL (bilirubin ≤1.5 x upper limit normal)
9. AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN and ≤ 5.0 ULN for subjects with liver metastases
10. Hemoglobin ≥ 7.5 g/dL and ≤ 13 g/dL
11. Absolute neutrophil count ≥1500/uL
12. Platelet count ≥ 75,000/ uL (>72 hours since prior platelet transfusion)
13. Corrected calcium within normal limits, previous hypercalcemia allowed
14. Females of childbearing potential must use a highly effective method of birth control for at least 28 days before starting study, during participation and at least 112 days following last dose of sotatercept.
15. Males must use latex condom or non-latex condom not made of (animal) membrane during any sexual contact with female of childbearing potential while participating in the study and for at least 112 days following the last dose of sotatercept, even if he has undergone successful vasectomy.

Exclusion Criteria:

1. History of thrombosis, deep vein thrombosis, pulmonary emboli, or embolic stroke AND have not been stable on anticoagulants within the past 6 months. Local central line thrombosis is allowed.
2. History of polycythemia
3. Uncontrolled hypertension (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg.)
4. History of severe allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or excipients in investigational product.
5. Current use of anti-cancer cytotoxic chemotherapeutic agents.
6. Major surgery within 30 days of Day 1 of trial.
7. Incomplete recovery or incomplete healing of wounds from previous surgery, as determined by treating Investigator.
8. Subjects with classification of 3 or higher heart failure as classified by the New York Heart Association (NYHA). Please see Appendix IV.
9. Women who are pregnant or breastfeeding or planning to become pregnant or breastfeed during the period of treatment and for 112 days following the last dose of sotatercept.
10. Treatment with another investigational drug or device within 28 days prior to Day 1, or if the half-life of the previous product is known, within 5 times the half-life of the investigational drug prior to dosing, whichever is longer.
11. Prior exposure to sotatercept.
12. Any significant medical condition, laboratory abnormality, or psychiatric illness that, as determined by the treating Investigator, would prevent the subject from participating in the study or providing written informed consent.
13. Any condition including the presence of laboratory abnormality that, as determined by the treating Investigator, places the subject at unacceptable risk if he/she were to participate in the study.
14. Known positive for human immunodeficiency virus (HIV)
15. Known positive for infectious hepatitis type C or active infectious hepatitis type B.
16. Any condition that, as determined by the treating Investigator, confounds the interpretation of data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Presence of biochemical bone turnover | Average of 3 months
  The presence of change in biochemical markers of bone turnover during treatment with sotatercept will be examined.

SECONDARY OUTCOMES:
Number of Adverse Events related to sotatercept | Average of 21 days
Bone marrow density | Average of 12 months
  Change in bone mineral density of the femoral neck, forearm and spine.
Change in biochemical myeloma markers | Average of 3 months
  The change in myeloma markers will be determined by quantifying immunoglobulins, SPEP, UPEP and free light chains.
Size of target bone lesions | Average of 6 months
  Measure the change in size of target bone lesions using x-ray of target skeletal lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Silbermann, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States